CLINICAL TRIAL: NCT06586216
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL STUDY TO ASSESS THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-07817883 IN ADULT PARTICIPANTS WITH RENAL IMPAIRMENT AND HEALTHY ADULT PARTICIPANTS WITH NORMAL RENAL FUNCTION
Brief Title: A Study to Learn How Renal Impairment Affects the Pharmacokinetics of PF-07817883.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C5091015
Record Dates: First submitted 2024-08-01; First posted 2024-09-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: Renal Impairment; COVID-19
MeSH Terms: conditions — COVID-19; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): No renal impairment
  Interventions: Drug: PF-07817883
- Cohort 2 (Experimental): Severe renal impairment
  Interventions: Drug: PF-07817883
- Cohort 3 (Experimental): Moderate renal impairment
  Interventions: Drug: PF-07817883

INTERVENTIONS:
Drug: PF-07817883 — Experimental

SUMMARY:
The purpose of the study is to learn about:

* how PF-07817883 is processed in the body of adult participants.
* the safety of PF-07817883.

These participants will have different levels of kidney function loss:

* moderate
* severe
* none or healthy Participants with moderate, severe or no loss of kidney function may be taken into one of 3 groups.

This study is seeking for participants who:

* are male or female of 18 to 90 years of age.
* have different levels of damage to kidney function or for one of the groups, no damage
* are willing to follow the requirements of the study including stay at clinic for 5 nights and 6 days.

About, 8 participants may be selected in groups 2 and 3. In group 1, around 8 to 12 participants may be selected. If participants agree to take part in the study, it may take up to 4 weeks to complete all the tests to confirm if they are fit to be in the study. If they seem to be fit for the study, participants will be admitted to a clinic research unit (CRU) at least 8 hours before dosing.

On Day 1, participants will receive a single amount of study medicine (Day 1). A series of blood samples will be collected before and after giving medicines. Participants will be discharged from the CRU on Day 5. A follow-up phone call (or CRU visit, if needed), will occur 28-35 days after taking the medicine. The whole study will last for a minimum of 5 weeks and a maximum of 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 (or the minimum age of consent in accordance with local regulations) to 90 years of age at screening.
* BMI of ≥16 kg/m2 and a total body weight >45 kg (99 lbs).
* Stable renal function, defined as the eGFR values obtained at the two screening visits should not be more than 25% different.

Exclusion Criteria:

* Positive test result for severe acute respiratory syndrome coronavirus 2 (SARS CoV 2) infection at the time of screening or Day -1.
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing at screening for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody (HCVAb). As an exception, a positive hepatitis B surface antibody (HBsAb) test due to hepatitis B vaccination is allowed.
* Renal transplant recipients.
* Any condition possibly affecting drug absorption

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-07817883 | Day 1 to Day 5
  Plasma PF-07817883 PK parameters
Area under the Plasma Concentration-time Profile from Time Zero to Extrapolated Infinite Time (AUCinf) | Day 1 to Day 5
  Plasma PF-07817883 PK parameters
Area under the Plasma Concentration-time Profile from Time Zero to the Time of the Last Quantifiable Concentration (AUClast) | Day 1 to Day 5
  Plasma PF-07817883 parameters

SECONDARY OUTCOMES:
Number of participants with Non-Serious Adverse Events (NSAE) | Screening to Day 35
  Safety Parameter
Number of participants with Treatment Emergent Adverse Events | Day 1 to Day 35
  Safety Parameter
Number of participants with Clinically Significant ECG Abnormalities | Day 1 to Day 5
Number of participants with Clinically Significant Abnormal Vital Signs | Day 1 to Day 5
Number of participants with Clinically Significant abnormal laboratory values. | Baseline to Day 5
Number of participants with Serious Adverse Events | Screening to Day 35
  Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091015